CLINICAL TRIAL: NCT00483132
Title: Study of Treatment High Risk and/or Low Risk Acute Lymphoblastic leukémia(ALL) Adults Stage III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GOELAL02
Record Dates: First submitted 2007-06-05; First posted 2007-06-06 (Estimated); Last update posted 2007-06-06 (Estimated); Status verified 2007-06

CONDITIONS: Leukemia, Lymphocytic, Acute
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Interferon alpha-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: interferon alpha 2a

SUMMARY:
Improved outcome of high risk lymphoblastic leukemia (ALL) with laite high dose therapy.

High dose versus conventional therapy for adult low risk T-ALL and Lymphoblastic lymphoma (LBL).

DETAILED DESCRIPTION:
Comparison between two autograf therapeutic strategies in high risk patients Ramdomised comparison between maintenance treatment with or not interferon alpha 2 a

ELIGIBILITY:
Inclusion Criteria

* ALL high risk or low risk or lymphoblastic lymphoma
* age 15-55 years old
* informed consent signed

Exclusion Criteria:

* patients previously treated with a chemotherapy or alpha-interferon
* ALL 3 (burkitt like)

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 1994-09; Study Completion 2002-04 (Actual)

PRIMARY OUTCOMES:
overall survival | time to death

SECONDARY OUTCOMES:
Efficacy of study treatments | time to end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Norbert IFRAH, Pr, Principal Investigator — French Innovative Leukemia Organisation; Noël MILPIED, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- INorbert IFRAH, Angers, Chu Angers, France

REFERENCES:
- [Result] Hunault M, Harousseau JL, Delain M, Truchan-Graczyk M, Cahn JY, Witz F, Lamy T, Pignon B, Jouet JP, Garidi R, Caillot D, Berthou C, Guyotat D, Sadoun A, Sotto JJ, Lioure B, Casassus P, Solal-Celigny P, Stalnikiewicz L, Audhuy B, Blanchet O, Baranger L, Bene MC, Ifrah N; GOELAMS (Groupe Ouest-Est des Leucemies Airgues et Maladies du Sang) Group. Better outcome of adult acute lymphoblastic leukemia after early genoidentical allogeneic bone marrow transplantation (BMT) than after late high-dose therapy and autologous BMT: a GOELAMS trial. Blood. 2004 Nov 15;104(10):3028-37. doi: 10.1182/blood-2003-10-3560. Epub 2004 Jul 15. PMID 15256423